CLINICAL TRIAL: NCT00224939
Title: Pre-ESRD Syndrome in High Risk African American Young Adults
Brief Title: Pre-ESRD Syndrome in High Risk African Americans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only apx 1/3 of enrolled subjects (signed consent) participated. Futility analysis to show primary endpoint
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DK 62714 (terminated)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Potassium Chloride

INTERVENTIONS:
Drug: Potassium Chloride

SUMMARY:
Evaluation of the dipping status of blood pressure (wether blood pressure decreases at night) and renal functional reserve and wether non-dippers (those whose blood pressure does not decrease at night) can be modulated to dippers with potassium treatment.

DETAILED DESCRIPTION:
Evaluation of the dipping status of blood pressure (wether blood pressure decreases at night) and renal functional reserve and wether non-dippers (those whose blood pressure does not decrease at night) can be modulated to dippers with potassium treatment.

ELIGIBILITY:
Inclusion Criteria: 18-35, healthy volunteers, African American

Exclusion Criteria: Active medical conditions, prescription drug therapy other than birth control

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2002-07; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Ripley, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States